CLINICAL TRIAL: NCT07090512
Title: Multimodal Ultrasound Assessment of Kidneys From Donation After Brain Death (DBD) to Predict the Risk Model of Early Postoperative Renal Insufficiency in Renal Transplantation
Brief Title: Multimodal Ultrasound in DBD Kidneys for Predicting Early Postoperative Renal Insufficiency Risk
Status: Recruiting | Type: Observational
Sponsor: Bei Wang (Other)
Responsible Party: Sponsor-Investigator, Bei Wang, Chief Physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2024(172)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Occurrence of Renal Dysfunction (GFR ≤ 60mL/(Min·1.73m2)) in Renal Transplant Recipients Within One Year After Kidney Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multimodal Ultrasound — Multimodal ultrasound data collection will be conducted on all organ donors meeting the research criteria.

SUMMARY:
The objective of this observational study is to investigate the multimodal ultrasound parameters of kidneys from brain-dead organ donors prior to donation, in order to construct a predictive model for assessing the risk of early transplant renal dysfunction after kidney transplantation in recipients.

The primary question this study aims to address is:

Can multimodal ultrasound data from brain-dead organ donor kidneys accurately predict early post-transplant renal dysfunction?

Ultrasonography, as a routine examination before organ donation, will be utilized, and the study results will be concluded within one year after participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Recipient Study Participants Age ≥18 years;

Underwent allogeneic kidney transplantation at this hospital;

Signed informed consent form.

Donor Study Participants Brain-deceased organ donors;

Completed organ donation at the First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province);

Brain death criteria:

Deep coma (with clear etiology and exclusion of reversible causes);

Absence of brainstem reflexes;

No spontaneous respiration;

Confirmed by at least two confirmatory tests (SLSEP, EEG, TCD), with re-evaluation 12 hours after the initial determination.

Standard Criteria Donor (SCD):

* Age 10-39 years;

  * Cause of death unrelated to cerebrovascular disease;

    * Serum creatinine <133 μmol/L;

      * No history of hypertension.

Expanded Criteria Donor (ECD):

* Age >60 years; OR

  ② Age 50-59 years with two of the following three criteria:
* Cause of death related to cerebrovascular disease;

  * Serum creatinine <133 μmol/L;

    * History of hypertension.

Signed informed consent form.

Exclusion Criteria:

* Recipient Study Participants Patients with multiple kidney transplants;

Patients with follow-up duration less than 1 year;

Patients experiencing irreversible loss of graft function due to postoperative complications (e.g., rejection, thrombosis, anastomotic stenosis, infection).

Donor Study Participants Severe primary renal diseases (e.g., hypertensive nephropathy, diabetic nephropathy, renal tumors);

Cases with unavailable ultrasound imaging data:

Excessive respiratory motion in donors;

Obesity or other factors affecting imaging quality.

Individuals with allergic predisposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Brain-deceased organ donors and their matched kidney transplant recipients at the First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province).
Sampling Method: Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
chronic allograft dysfunction | Development of chronic allograft dysfunction within one year following kidney transplantation.
  Occurrence of chronic allograft dysfunction (GFR ≤ 60mL/(min·1.73m2)) in renal transplant recipients within one year after kidney transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China